CLINICAL TRIAL: NCT04413383
Title: Do Patients Undergoing Dermatologic Surgery Prefer the Use of Traditional Curved Iris Scissors or the Wuennenberg Modified Curved Iris Scissors?
Brief Title: Use of Traditional Curved Iris Scissors or the Wuennenberg Modified Curved Iris Scissors for Skin Surgery
Acronym: TISMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, John Wuennenberg, Resident Physician, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023744
Record Dates: First submitted 2020-05-19; First posted 2020-06-02 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Traditional Curved Iris Scissors (Active Comparator): The traditional curved Iris scissors are used to during the dermatologic surgery. Patients complete a survey after the surgery on sights, sounds and smells experienced during the procedure.
  Interventions: Other: Traditional Curved Iris Scissors
- Modified Curved Iris Scissors (Experimental): The Wuennenberg modified curved Iris scissors are used during the dermatologic surgery.
  Patients complete a survey after the surgery on sights, sounds and smells experienced during the procedure.
  Interventions: Other: Wuennenberg Modified Curved Iris Scissors
- Comparative Experience (Other): Both the traditional and modified curved Iris scissors are used and patients are asked which they prefer. Patients complete a survey after the surgery on sights, sounds and smells experienced during the procedure.
  Interventions: Other: Comparative Experience of Traditional and Wuennenberg Modified Curved Iris Scissors

INTERVENTIONS:
Other: Traditional Curved Iris Scissors — Aesculap Curved Iris Scissors
  Other Names: Curved Iris Scissors
  Arms: Traditional Curved Iris Scissors
Other: Wuennenberg Modified Curved Iris Scissors — Modified Silent Curved Iris Scissors
  Other Names: Modified Curved Iris Scissors
  Arms: Modified Curved Iris Scissors
Other: Comparative Experience of Traditional and Wuennenberg Modified Curved Iris Scissors — Patients experience both types of scissors
  Other Names: Comparative Experience
  Arms: Comparative Experience

SUMMARY:
Every year thousands of dermatologic surgery procedures are performed at the University of Missouri Department of Dermatology, including Mohs Micrographic Surgery (MMS), Excisions, and biopsies. Surgery is known to cause anxiety for patients and with these procedures performed under local anesthetic on awake patients', the sights, sounds, and smells experienced during the procedure can lead to an increase in their anxiety or affect their overall perception of the experience. From performing and assisting with dermatologic surgery the noise associated with the use of the traditional curved Iris scissors provokes an increase in patient awareness to the procedure resulting in increased anxiety, triggering of the vasovagal response, and expressions of annoyance by the patient. However, the modified curved Iris scissors make almost no noise. The Investigators hypothesize that if patients were given the comparative experience of both types of curved Iris scissors during dermatologic surgery, then they will choose the modified curved Iris scissors because the lack of noise will be perceived as more pleasant experience. Our objective is to perform a prospective, single blinded, randomized controlled trial to determine how the noise of traditional curved Iris scissors vs the silent Wuennenberg modified curved Iris scissors affects patients during dermatologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* non-pregnant
* patients being treated with Mohs micrographic surgery or excision on the head and neck

Exclusion Criteria:

* Patients not meeting above inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Extent that patient notices curved Iris scissors | 3 to 8 hours (length of the patients Mohs Surgery)
  Questionnaire with an ordinal scale from 1 to 10 to assess the extent that patient notices the use of the curved iris scissors.
Extent that patient is bothered by the curved Iris scissors | 3 to 8 hours (length of the patients Mohs Surgery)
  Questionnaire with an ordinal scale from 1 to 10 to assess the extent that patient is bothered by the curved iris scissors.
Patients Preference of curved Iris scissor | 3 to 8 hours (length of the patients Mohs Surgery)
  Patient is asked during the procedure if they prefer "1," surgeon uses the traditional curved Iris scissors, or "2" and the surgeon uses the Wuennenberg modified curved Iris scissors. The patient indicates their preference by responding "1 or 2." After the procedure the patient completes a questionnaire with an ordinal scale from 1 to 10 to assess the extent that patient notices and is bothered by the curved iris scissors.

CONTACTS AND LOCATIONS:
Overall Officials: John P Wuennenberg, MD, Principal Investigator — University of Missouri-Columbia Dermatology
Locations (1):
- UPMB, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No